CLINICAL TRIAL: NCT04709042
Title: Acquisition of Objective Data During Transapical Neochordae Implantation
Acronym: TENSCHORD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no more medical device implantation
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL19_1034; ID-RCB (Other: 2020-A02208-31)
Record Dates: First submitted 2021-01-11; First posted 2021-01-14 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Mitral Valve Insufficiency; Mitral Regurgitation
Keywords: Primary Mitral Regurgitation; Mitral Valve repair; Heart Surgery; Neochord DS1000; Intraoperative Chordal Tension; Tension Measurement; Cardiac Magnetic Resonance Imaging; Postoperative echocardiographic evaluation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chordal tension measurement and cardiac Magnetic Resonance Imaging (Experimental): All patient candidates for NeoChord implantation according to the standard of care will be considered for inclusion in this clinical study. Chordal tension measurement will be performed during Neochord implantation. Moreover, all patients will undergo cardiac Magnetic Resonance Imaging (MRI) exam before the surgery, as well as at 3 months follow-up.
  Interventions: Procedure: Chordal tension measurement; Other: Cardiac Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Procedure: Chordal tension measurement — The chordal tension measurement will be performed during surgery. The neochordae are connected to the measuring device through "crocodile" clips (e.g. machine-patient interface).We start to apply traction on the chordae that is in the center of the flailing area thanks to a millimeter screw and under TEE control. After obtaining a stable tension (plateau value), the other chordae are then tracked, one at a time, with an individual screw. When we achieve an equivalent tension on all chordae, a traction on all chordae is applied thanks to the principal screw under TEE control until obtaining a perfect coaptation. When the correction is optimal (good echocardiographic result, chordal tension low and equally spread on each chordae), the measurements are then stopped, and the chordae are fixed at the apex of the left ventricle at the optimal length.
Other: Cardiac Magnetic Resonance Imaging (MRI) — Patients will undergo 2 MRI exams: 1 MRI before surgical intervention (maximum 21 days before) and 1 MRI three months after surgery (+/- 14 days), with intravenous administration of gadolinium.

SUMMARY:
Mitral Valve repair (MVr) is the gold standard treatment for primary Mitral Regurgitation. Implantation of artificial Gore-Tex chordae (or neochordae implantation) is often used for MVr.

The NeoChord DS1000 (NeoChord Inc., Minneapolis, USA) is a device designed to deploy neochordae through transapical access in a beating heart and without cardiopulmonary bypass. NeoChord System is CE marked and therefore authorized for use in Europe. Procedure is conducted under 3D transesophageal echocardiography (TEE) guidance. The device is introduced through the apex of the left ventricular (LV) and the prolapsed leaflet is grabbed and harpooned.

The neochordae are thus stretched between the valve and the LV apex. Neochordae length can be precisely adapted to restore a normal coaptation, to treat the regurgitation.

Recently, the principal investigator's teams (heart surgery department at Hospices Civils de Lyon and Laboratoire de Génie Electrique et Ferromagnétique lab at Institut National des Sciences Appliquées (INSA) de Lyon, France) created a platform allowing the measurement of the tension applied on neochordae during a NeoChord procedure. A dedicated protocol was designed and approved by the ethical committee of the French Society of Cardiology. The measurement was performed in 7 patients. This preliminary study shows that the technic is safe. It also suggests that chordal tension might be correlated to the quality of MVr: the sub-valvular apparatus appears to be in a low stress state when the structure and the function of the valve are restored.

These first findings raise new questions:

1. The mechanism involved in the changes in tensions during chordal length adjustment cannot be understood with current standard medical imaging tools. Numerical simulation technologies could bring physical data in order to approach physical phenomenon underlying these findings.
2. Novel chordal tension measurement tools could lead to a change in current paradigm enabling a MVr based on objective data measurement, instead of sole morphological analysis. Prognostic value of chordal tension must be studied through a larger clinical study and a systematic protocol.

A large consortium involving physicians and scientists has been created to address those questions, and a large national funding has been raised to fulfil our objectives over a 4 years period (SIMR project). The present clinical study is the core of this large project.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old)
* Patient candidate for NeoChord procedure after validation by the local Heart-Team

  * severe symptomatic MR due to a posterior prolapses, involving mainly the P2 segment (with a variable extension on P1 or P3, but never involving the commissures or the anterior leaflet). Also, a LAI (leaflet to annulus index) >1,25 will be required.
  * and considered as high-risk for conventional surgery (mainly because of frailty) after selection by our heart team.
* Patient who has provided his written informed consent to participate in the study
* Patient affiliated to a social health insurance.

Exclusion Criteria:

* Patient with contraindication for NeoChord technic including:

  * Patient with secondary MR
  * LV dilatation with initial tethering
  * Central component to regurgitant jet
  * Calcified leaflets segments.
* Patient with contraindication for Cardiovascular Magnetic Resonance (CMR) imaging:

  * Patients without sinus rhythm
  * Regular MRI contraindications (e.g. a pacemaker, defibrillator or metallic (ferromagnetic) body, a known allergy to gadolinium)
  * Contraindication for Gadolinium infusion : glomerular filtration rate (GFR) <30 ml / min
* Patient unable to understand the purpose of the study
* Patient participating in another trial that would interfere with this study
* Female patient who is pregnant or lactating
* Patients under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Correlate intraoperative chordal tension and postoperative echocardiographic mitral valve repair success (defined as mitral regurgitation (MR) ≤2+) | Day 0
  Correlation between intraoperative chordal tension (measured in mmHg) and postoperative echocardiographic mitral valve repair success (defined as mitral regurgitation (MR) ≤2+)
Correlate intraoperative chordal tension and postoperative echocardiographic mitral valve repair success (defined as mitral regurgitation (MR) ≤2+) | 1 month after surgery
  Correlation between intraoperative chordal tension (measured in mmHg) and postoperative echocardiographic mitral valve repair success (defined as mitral regurgitation (MR) ≤2+)
Correlate intraoperative chordal tension and postoperative echocardiographic mitral valve repair success (defined as mitral regurgitation (MR) ≤2+) | 12 months after surgery
  Correlation between intraoperative chordal tension (measured in mmHg) and postoperative echocardiographic mitral valve repair success (defined as mitral regurgitation (MR) ≤2+)

SECONDARY OUTCOMES:
Duration of procedure in minutes | Day 0
  Intraoperative safety is assessed by procedure duration in minutes (defined as skin incision to skin closure)
Number of adverse events (AEs) and serious adverse events (SAEs) | 12 months
  Post-operative safety is assessed by occurrence of adverse events (AEs) and serious adverse events (SAEs) at each of the follow-up times
Duration of hospitalization | From the end of surgery (Day 0) to discharge from hospital (Day 15)
  Post-operative safety is assessed by duration of hospitalization
Number of patients with mitral regurgitation (MR) > 2+ | 1 month after surgery
  Mitral regurgitation is assessed by echocardiographic exam
Number of patients with mitral regurgitation (MR) > 2+ | 12 months after surgery
  Mitral regurgitation is assessed by echocardiographic exam
Number of rehospitalization for heart failure and mitral valve reoperation | 1 month after surgery
  Freedom from rehospitalization for heart failure and Mitral valve reoperation free survival
Number of rehospitalization for heart failure and mitral valve reoperation | 3 months after surgery
  Freedom from rehospitalization for heart failure and Mitral valve reoperation free survival
Number of rehospitalization for heart failure and mitral valve reoperation | 12 months after surgery
  Freedom from rehospitalization for heart failure and Mitral valve reoperation free survival
New York Heart Association (NYHA) score | Inclusion
  Change in functional evaluation is assessed by NYHA functional classification of heart failure. It is based on symptom severity and the amount of exertion needed to provoke symptoms. NYHA heart failure classes are as follows : Class I No limitation of physical activity, Class II Slight limitation of physical activity, in which ordinary physical activity leads to fatigue, palpitation, or dyspnea; the person is comfortable at rest, Class III Marked limitation of physical activity, in which less-than-ordinary activity results in fatigue, palpitation, or dyspnea; the person is comfortable at rest and Class IV Inability to carry on any physical activity without discomfort but also symptoms of heart failure at rest, with increased discomfort if any physical activity is undertaken.
New York Heart Association (NYHA) score | Discharge from hospital (Day 15)
  Change in functional evaluation is assessed by NYHA functional classification of heart failure. It is based on symptom severity and the amount of exertion needed to provoke symptoms. NYHA heart failure classes are as follows : Class I No limitation of physical activity, Class II Slight limitation of physical activity, in which ordinary physical activity leads to fatigue, palpitation, or dyspnea; the person is comfortable at rest, Class III Marked limitation of physical activity, in which less-than-ordinary activity results in fatigue, palpitation, or dyspnea; the person is comfortable at rest and Class IV Inability to carry on any physical activity without discomfort but also symptoms of heart failure at rest, with increased discomfort if any physical activity is undertaken.
New York Heart Association (NYHA) score | 1 month after surgery
  Change in functional evaluation is assessed by NYHA functional classification of heart failure. It is based on symptom severity and the amount of exertion needed to provoke symptoms. NYHA heart failure classes are as follows : Class I No limitation of physical activity, Class II Slight limitation of physical activity, in which ordinary physical activity leads to fatigue, palpitation, or dyspnea; the person is comfortable at rest, Class III Marked limitation of physical activity, in which less-than-ordinary activity results in fatigue, palpitation, or dyspnea; the person is comfortable at rest and Class IV Inability to carry on any physical activity without discomfort but also symptoms of heart failure at rest, with increased discomfort if any physical activity is undertaken.
New York Heart Association (NYHA) score | 3 months after surgery
  Change in functional evaluation is assessed by NYHA functional classification of heart failure. It is based on symptom severity and the amount of exertion needed to provoke symptoms. NYHA heart failure classes are as follows : Class I No limitation of physical activity, Class II Slight limitation of physical activity, in which ordinary physical activity leads to fatigue, palpitation, or dyspnea; the person is comfortable at rest, Class III Marked limitation of physical activity, in which less-than-ordinary activity results in fatigue, palpitation, or dyspnea; the person is comfortable at rest and Class IV Inability to carry on any physical activity without discomfort but also symptoms of heart failure at rest, with increased discomfort if any physical activity is undertaken.
New York Heart Association (NYHA) score | 12 months after surgery
  Change in functional evaluation is assessed by NYHA functional classification of heart failure. It is based on symptom severity and the amount of exertion needed to provoke symptoms. NYHA heart failure classes are as follows : Class I No limitation of physical activity, Class II Slight limitation of physical activity, in which ordinary physical activity leads to fatigue, palpitation, or dyspnea; the person is comfortable at rest, Class III Marked limitation of physical activity, in which less-than-ordinary activity results in fatigue, palpitation, or dyspnea; the person is comfortable at rest and Class IV Inability to carry on any physical activity without discomfort but also symptoms of heart failure at rest, with increased discomfort if any physical activity is undertaken.
The 3-level version of EQ-5D (EQ-5D-3L) health status score (quality of life score) | Inclusion
  The EQ-5D-3L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
The 3-level version of EQ-5D (EQ-5D-3L) health status score (quality of life score) | Discharge from hospital (Day 15)
  The EQ-5D-3L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
The 3-level version of EQ-5D (EQ-5D-3L) health status score (quality of life score) | 1 month after surgery
  The EQ-5D-3L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
The 3-level version of EQ-5D (EQ-5D-3L) health status score (quality of life score) | 3 months after surgery
  The EQ-5D-3L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
The 3-level version of EQ-5D (EQ-5D-3L) health status score (quality of life score) | 12 months after surgery
  The EQ-5D-3L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Left ventricular volumes and function quantification | Inclusion
  Left ventricular volumes and function quantification are assessed by Cardiac Magnetic Resonance Imaging (MRI)
Left ventricular volumes and function quantification | 3 months after surgery
  Left ventricular volumes and function quantification are assessed by Cardiac Magnetic Resonance Imaging (MRI)
Number of left ventricular tissue fibrosis | Inclusion
  Left ventricular tissue fibrosis are assessed by Cardiac Magnetic Resonance Imaging (MRI)
Number of left ventricular tissue fibrosis | 3 months after surgery
  Left ventricular tissue fibrosis are assessed by Cardiac Magnetic Resonance Imaging (MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel GRINBERG, MD, Principal Investigator — Hôpital Pneumologique et Cardiovasculaire Louis Pradel

REFERENCES:
- [Result] Grinberg D, Cottinet PJ, Thivolet S, Audigier D, Capsal JF, Le MQ, Obadia JF. Measuring chordae tension during transapical neochordae implantation: Toward understanding objective consequences of mitral valve repair. J Thorac Cardiovasc Surg. 2019 Sep;158(3):746-755. doi: 10.1016/j.jtcvs.2018.10.029. Epub 2018 Oct 17. PMID 30454983